CLINICAL TRIAL: NCT03981705
Title: Assessment of Complete Pathologic Response After Neoadjuvant Chemotherapy for Breast Cancer
Status: Completed | Type: Observational
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 2018NTLS176
Record Dates: First submitted 2019-06-07; First posted 2019-06-11 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: TN ER-/PR-/HER2- Breast Cancer; Triple Negative Breast Cancer; HER2-positive Breast Cancer; ERany/PRany/HER2+ Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Standard Trimodality Breast Imaging — Standard breast imaging with or without core needle biopsy after neoadjuvant chemotherapy (NAC).

SUMMARY:
This is a feasibility study to gain preliminary information regarding whether breast imaging with or without a core needle biopsy after neoadjuvant chemotherapy (NAC) but before surgery can accurately predict complete pathologic response (pCR) in women with triple negative or HER2- positive breast cancer. pCR is defined as having no residual invasive breast cancer or ductal carcinoma in situ.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven triple negative (TN) (ER-/PR-/HER2-) or HER2 positive (ERany/PRany/HER2+) breast cancer for which neoadjuvant chemotherapy is planned
* A biopsy clip placed at the time of diagnostic biopsy
* 18 years of age or older
* Must be able to read and write in English due to the importance of survey (questionnaire) completion to meet the study's endpoint - this is justified as there is no individual benefit to study participation
* Able to provide written consent prior to any research related activities

Exclusion Criteria:

* Stage IV breast cancer
* T4 breast cancer
* Previous ipsilateral breast cancer
* Any contraindication for undergoing a contrast-enhanced breast MRI and/or the breast biopsy between chemotherapy and surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study entry is open to women 18 years of age and older regardless of race or ethnic background. While there will be every effort to seek out and include minority patients, the patient population is expected reflect those at the University of Minnesota with triple negative or HER2+ breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2024-11-26 (Actual)

PRIMARY OUTCOMES:
Complete Pathologic Response (pCR) | 6 Months Post Surgery
  The primary aim of this feasibility study is to determine whether breast imaging with or without core needle biopsy after neoadjuvant chemotherapy (NAC) can accurately predict complete pathologic response (pCR) in women with biopsyproven triple negative or HER2+ breast cancer.

SECONDARY OUTCOMES:
Complications and Side Effects of the Needle Biopsy Procedure after NAC | 6 Months Post Surgery
  Incidence of Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Todd Tuttle, MD, MS, Principal Investigator — Department of Surgery, University of Minnesota
Locations (1):
- University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota, United States